CLINICAL TRIAL: NCT05207826
Title: Determining the Most Appropriate Time to Evaluate Detrusor Activity Recovery in Acute Traumatic Spinal Cord Injuries
Brief Title: Detrusor Activity Recovery in Acute Traumatic Spinal Cord Injuries
Status: Withdrawn | Type: Observational
Why Stopped: Cancelled to conduct study on similar but more appropriate topics
Sponsor: Pusan National University Yangsan Hospital (Other)
Collaborators: Coloplast A/S (Industry)
Responsible Party: Principal Investigator, Sungchul Huh, Assistant professor, Pusan National University Yangsan Hospital
Other Study IDs: DRASS
Record Dates: First submitted 2021-12-28; First posted 2022-01-26 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Spinal Cord Injuries; Neurogenic Bladder; Spinal Shock
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cystometrogram — Serial cystometrogram every 3 days for acute traumatic spinal cord injured patients

SUMMARY:
Determining the most appropriate time to evaluate detrusor activity in urodynamic studies for both traumatic and non-traumatic spinal cord injuries

DETAILED DESCRIPTION:
The detrusor activity in the acute phase of the spinal cord injury changes with the development of the spinal shock. Spinal shock is a phase of areflexic phase after the spinal cord injury that is primarily influenced by the severity of the injury and the neurological level of injury. Detrusor activity shows areflexic in the spinal shock phase, followed by a return of detrusor activity at the end of the spinal shock.

There was no recent study to provide evidence of an appropriate time to assess detrusor muscle activity through urodynamic studies. There were only a few limited studies on detrusor activity following spinal cord injury from 1960 to 1970. However, when the urodynamic study should be performed is still controversial.

Knowing the patterns of detrusor activity following spinal cord injuries is critical to determining the appropriate timing for intermittent catheterization, which is the standard emptying method of choice. If clinicians fail to understand true detrusor activity as early as possible, the patient will suffer from unnecessary indwelling catheter voiding, resulting in impaired quality of life in the acute phase.

ELIGIBILITY:
Inclusion Criteria:

* Acute onset suprasacral spinal cord injury with both traumatic and non-traumatic causes within the first 15 days after spinal cord injury(very acute phase of SCI according to European Multicenter Study about SCI : the first 15 d (very acute), between 16-40 d (acute I), and 3 mo (acute II), 6 mo (acute III), and 12 mo (chronic) after SCI)
* Age older than 18
* Inpatient
* Patients with spinal cord injuries who initially keep the indwelling catheter
* Patients with or without spinal shock

Exclusion Criteria:

nstable vital sign (using Inotropics or vasopressors or antiarrhythmic agents)

* Current urinary tract infection
* Agitated behavior (Richmond Agitation and Sedation Scale of +2 to +4)
* Decreased mentality (RASS of -2 to -5)
* Concomitant sacral lesions (Ex. Sacral fracture, pelvic bone fracture, urologic trauma)
* Concomitant supraspinal lesions (Ex. Traumatic brain injury, old stroke, Parkinson disease)
* Uncontrolled DM
* Medical history of lower urinary tract dysfunction (Ex. BPH, Malignancy)
* Uncontrlled autonomic dysreflexia (In case of autonomic dysreflexia, defined according to ISAFSCI (International Standards to document remaining Autonomic Function after SCI) as an increase in systolic blood pressure 20 mm Hg or greater from baseline

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute traumatic spinal cord injuries
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Detrusor activity recovery | Every 3 days in spinal shock phase (up to 3 months)
  Pressure change (Detrusor pressure change in filling cystometrogram)

SECONDARY OUTCOMES:
Reflexes | Every 3 days in spinal shock phase (up to 3 months)
  Superficial reflex and pathologic reflex (Cremasteric reflex, Dartos reflex, BC reflex, anal reflex, Babinski reflex, delayed plantar reflex)

CONTACTS AND LOCATIONS:
Overall Officials: Sungchul Huh, PhD, Principal Investigator — Pusan National University Yangsan Hospital

IPD SHARING:
Plan to Share IPD: No